CLINICAL TRIAL: NCT00998777
Title: The Effect of a 6-week Shoulder Strengthening Program on Scapular Kinematics and Shoulder Strength in Division I Collegiate Swimmers
Brief Title: Shoulder Injury Prevention Program in Swimmers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SwimmersShoulder
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Shoulder Injury
Keywords: tubing program; shoulder strengthening; injury prevention
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shoulder Strengthening (Experimental): The shoulder strengthening program is a 6-week intervention aimed to improve shoulder and scapular stabilizer strength and scapular kinematics. The program includes 10 exercises: shoulder flexion, Ys,Ts,Ws, Throwing Acceleration, Throwing Deceleration, Low Rows, Dynamic Hug, IR @ 90, and ER @ 90. The program also includes 2 stretches: sleeper stretch and corner stretch.
  Interventions: Procedure: Shoulder Strengthening

INTERVENTIONS:
Procedure: Shoulder Strengthening — The intervention program is a 6 week shoulder and scapular stabilizer strengthening program that is performed 3 times per week. The program includes 10 exercises that are performed with Theraband rubber tubing and 2 stretches. The exercises are: shoulder flexion, Ys, Ts, Ws, IR @ 90, ER @ 90, Throwing acceleration, Throwing deceleration, dynamic hug, and low rows. The stretches include the sleeper stretch and the corner stretch.
  Other Names: Shoulder injury prevention, tubing program for athletes

SUMMARY:
The primary purpose of this study is to assess changes in shoulder muscle strength, shoulder movement, shoulder flexibility, muscle thickness, upper arm torsion angle, and subacromial width (space where the rotator cuff muscle passes through) after completing a 6-week shoulder strengthening and stretching program in division I collegiate swimmers. The result of this study may demonstrate the effectiveness of a strengthening and stretching program to positively influence factors that have been associated with pain and injury in division I collegiate swimmers and indicate the need to implement this program for the entire team. Following a 6-week strengthening and stretching program, it is believed that scapular kinematics, shoulder flexibility, and shoulder and scapular stabilizer strength will be improved compared to control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included in the study if they meet the following criteria:

  * NCAA division I swimmers
  * Participate in swimming for at least 30 minutes per day for 4 days per week.
  * Participate in all team weight lifting sessions.
  * Complete 15 of the 18 training sessions if the subject is placed in the treatment group.

Exclusion Criteria:

* Subjects will be excluded from the study if:

  * They are currently being treated for shoulder pain
  * They develop shoulder pain during the course of the intervention program

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Shoulder and Scapular Stabilizer Strength | Measured pre and post test

SECONDARY OUTCOMES:
Scapular Kinematics | Measured pre and post test
Shoulder ROM | Measured pre and post test
Postural Assessment | Measured pre and post test
Width of subacromial space | Measured pre and post test

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hibberd, Principal Investigator — UNC-Chapel Hill; Joseph B Myers, PhD, ATC, Study Director — UNC- Chapel Hill
Locations (1):
- Dean E. Smith Center, Chapel Hill, North Carolina, United States